# Title:

# ELECTROPHYSIOLOGICAL STUDIES OF INDUCED FORWARD HEAD POSITION AND HAND USE OF MOBIL PHONE

NCT: not yet assigned

Document Date: 12/11/2019

# FACULTY OF PHYSICAL THERAPY APPLICATION FOR ETHICAL REVIEW

# **NOTES:**

- Answers to questions must be entered in the space provided.
- An electronic version of the completed form should be submitted to the Research Ethics

  Officer, at the following email address: <a href="mailto:...ethical@pt.cu.edu.eg.....">...ethical@pt.cu.edu.eg.....</a>. Please **do not** submit paper copies.
- If you have any queries about the form, please address them to the Research Ethics Team

# FACULTY OF PHYSICAL THERAPY APPLICATION FOR ETHICAL REVIEW

| OFFICE USE ONLY: |
|------------------|
| Application No: |
| Date Received: |

| 1 | TIT | ΊF | OF | PR | OF | 20 | LΔ: |
|----|-----|----|----|--------------|----|----|-----|
| 1. | | | UГ | $\mathbf{r}$ | VГ | - | ᅭ |

| ELECTROPHYSIOLOGICAL STUDIES OF INDUCED FORWARD | <b>HEAD POSITION AND HAN</b> | D |
|---|---|---|
| USE OF MOBIL PHONE | | |

| 2. THIS | PROP | OSAL I | S: |
|---------|------|--------|----|
|---------|------|--------|----|

| Physical Therapy Staff Research Propo | sal 🗌 | | |
|---|---|---|---|
| Physical Therapy Postgraduate Research (PGR ☐ student Proposal √ ☐ | | | |
| | Master <sup>□</sup> | Doctoral $\sqrt{}$ | Other |
| Other Please specify): | | | |

# 3. INVESTIGATORS

# a) PLEASE GIVE DETAILS OF Student (FOR PGR STUDENT PROPOSAL) or first author for staff Research Proposal

| Name: Title / first name / family name | Karim sami ibrahim |
|---|---|
| Highest qualification & position held: | MSc. Of Pediatric Physical Therapy, Assistant Lecturer at MTI University |
| Department/ Faculty/ University Telephone: Email address: | Pediatrics/Physical Therapy/MTI university |
| | +2 01124252525 |
| | Karim_elsaharty25@yahoo.com |

# a) PLEASE GIVE DETAILS OF ANY CO-SUPERVISORS OR CO-INVESTIGATORS (FOR PGR STUDENT PROPOSAL) or co- first author for staff Research Proposal b)

| Name: Title / first name / family name | Prof. AMIRA EL-TOHAMY |
|---|---|
| Highest qualification & position held: | Professor |
| Department/ Faculty/ University Telephone: | Pediatrics/Physical Therapy/ Cairo University |
| Email address: | |
| | amiraeltahamy@yahoo.com |
| Name: Title / first name / family name | Ass.Prof. walaaabdelhakeem |
| Highest qualification & position held: | Assistant Professor |
| Department/ Faculty/ University Telephone: | Pediatrics/Physical Therapy/ Cairo University |
| Email address: | |
| | Walaa_abdelhakim@gmail.com |

| Name: Title / first name / family name Highest qualification & position held: Department/ Faculty/ University Telephone: | DR. MOHAMED HAMED RASHAD |
|---|---|
| | Lecturer of Neurology |
| | Pediatrics/Medicine/ Cairo University |
| Email address: | |

# 4. SUMMARY OF PROPOSAL

To compare between forward head position and hand use of mobile phone on conduction velocity of upper limb nerves

# **PURPOSE:**

- -To compare between forward head position and hand use of mobile phone on conduction velocity of upper limb nerves
- -To investigate the F responses of upper limbs nerves.
- -To investigate the compound muscle action potential (CMAP) amplitudes of median nerves

## **BACKGROUND:**

Forward head position may affect the cervical nerve root so it can also affect nerve conduction velocity due to continues stretch on nerves, also the over use of smart phone by hand may be affected the hand nerves, so this study determine which one of them has more influence than the other.

If the forward head position has the worst effect on the upper limb nerves we must avoid the incorrect position of the head to avoid stretch and compression of the nerves.

## **HYPOTHESES:**

-There are no statistical difference between forward head position and hand use of mobile phone on conduction velocity of the nerves of upper limb.

# **RESEARCH QUESTION:**

| ls there a | correlation | between ' | forward | head | position | and | hand | use | of r | nobile | phone | on |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| electrophy | siological p | oarameter | s of upp | er lim | b nerves | s? | | | | | | |

# 5. CONDUCT OF PROJECT

# Please give a description of the research methodology that will be used

| potential |
|---|
| 2- Soft collar Will used to fixed the craniovertebral angle during used mobile phone |
| 3- Universal goniometer Will used to measure craniovertebral angle |

# 6. PARTICIPANTS AS THE SUBJECTS OF THE RESEARCH

Describe the number of participants and important characteristics (such as age, gender, intellectual ability etc.). Specify any inclusion/exclusion criteria to be used.

Normal three hundred thirty five of both genders will participate in this study, Their ages range from 14-18 years, Not rolled on any regular athletic activity

Note: Attach a copy of any poster(s), advertisement(s) or letter(s) to be used for recruitment.

Inclusion criteria:

Their ages range from 14-18 years.

Not rolled on any regular athletic activity

-Exclusion criteria:

Individual with neck pain

Congenital deformity for upper limb

Peripheral neuropathy due to diabetes mellitus type I

Rheumatoid arthritis

History of surgical intervention at nerves of the upper extremity

# 8. CONSENT

Describe the process that the investigator(s) will be using to obtain valid consent. If consent is not to be obtained explain why. If the participants are minors or for other reasons are not competent to consent, describe the proposed alternate source of consent, including any permission / information letter to be provided to the person(s) providing the consent.

| I am freely and voluntarily consent to participate in a research program under the direction of M.Sc. |
|---|
| A thorough description of the procedure has been explained and I understand that I may withdraw r consent and discontinue participation in this research at any time without prejudice to me. Date Participant |
| Note: Attach a copy of the Consent Form, Participant Information Sheet (if applicable). |
| PARTICIPANT WITHDRAWAL |
| a) Describe how the participants will be informed of their right to withdraw from the project. |
| They can withdraw at anytime without prejudice to them as mention in signed consent. |
| b) Explain any consequences for the participant of withdrawing from the study and indicate what |
| will be done with the participant's data if they withdraw. |
| No consequences will take place. They have the utmost freedom. |
| . 15 55554.5555 Hill take place. They have the different fooders. |

# 9. CONFIDENTIALITY

| a) | Will all participants be anonymous? | Yes √ □ | No 🖳 | |
|----|-------------------------------------------|-----------------|------|---|
| b) | Will all data be treated as confidential? | Yes $\sqrt{\ }$ | No 💾 | Ц |

Note: Participants' identity/data will be confidential if an assigned ID code or number is used, but it will not be anonymous. Anonymous data cannot be traced back to an individual participant.

# 10. SIGNIFICANCE/BENEFITS

Outline the potential significance and/or benefits of the research

Delay in the treatment of extended Erb's palsy may result in substantial and chronic impairment due to many causes. One of the causes is the imbalance between the recovery of elbow lexors and elbow extensors where the latter will be delayed. This study will determine if a debilitating tightness and contracture (elbow flexion) can be prevented using the kinesiology tape in infants with Extended Erb's Palsy.

# **11. RISKS**

Outline any potential risks to **INDIVIDUALS**, including research staff, research participants, other individuals not involved in the research and the measures that will be taken to minimise any risks and the procedures to be adopted in the event of mishap

Risk of Infection: minimizing the risk through adequate sterilization of the treated areas during evaluation and treatment.

# 12. DECLARATION BY APPLICANTS

I submit this application on the basis that the information it contains is confidential and will be used by the Faculty of Physical Therapy for the purposes of ethical review and monitoring of the research project described herein, and to satisfy reporting requirements to regulatory bodies. The information will not be used for any other purpose without my prior consent.

# I declare that:

- The information in this form together with any accompanying information is complete and correct to the best of my knowledge and belief and I take full responsibility for it.
- I will report any changes affecting the ethical aspects of the project to the Faculty of Physical Therapy Research Ethics Officer.
- I will report any adverse or unforeseen events which occur to the relevant Ethics Committee via the Faculty of Physical Therapy Research Ethics Officer.

| Name of Principal investigator/project supervisor: | Karim sami ibrahim |
|----------------------------------------------------|-----------------------|
| | Prof. Amera El-Tohamy |
| Date: | 12 of novamber, 2019 |

# **Preflight Results**

# **Document Overview**

# **Preflight Information**

Title: Profile: Convert to PDF/A-1b

Author: El Khatib, Yehia (elkhatib) Version: Qoppa jPDFPreflight v2020R2.00

Creator: Microsoft® Word 2010 Date: Sep 14, 2020 7:25:59 AM

Producer: Microsoft® Word 2010

Legend: (X) - Can NOT be fixed by PDF/A-1b conversion.

(!X) - Could be fixed by PDF/A-1b conversion. User chose to be warned in PDF/A settings.

# Page 1 Results

- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman, Bold is not embedded. Font Times New Roman, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman, Bold is not embedded. Font Times New Roman, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman,Bold is not embedded. Font Times New Roman,Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman, Bold is not embedded. Font Times New Roman, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman,Bold is not embedded. Font Times New Roman,Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman,Bold is not embedded. Font Times New Roman,Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman, Bold is not embedded. Font Times New Roman, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman, Bold is not embedded. Font Times New Roman, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman, Bold is not embedded. Font Times New Roman, Bold can not be embedded because: Could not find matching font to embed


- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed


- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed 6 more not displayed

## Page 2 Results

- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed


- (X) Font Arial,Bold is not embedded. Font Arial,Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed 3 more not displayed


- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Italic is not embedded. Font Arial, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Italic is not embedded. Font Arial, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed


- (X) Font Arial,Bold is not embedded. Font Arial,Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman, Italic is not embedded. Font Times New Roman, Italic can not be embedded because: Could not find matching font to embed


- (X) Font Arial,Bold is not embedded. Font Arial,Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman, Italic is not embedded. Font Times New Roman, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Italic is not embedded. Font Arial, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Italic is not embedded. Font Arial, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed 29 more not displayed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed 53 more not displayed


- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed


- (X) Font Arial,Bold is not embedded. Font Arial,Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed 24 more not displayed


- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed


- (X) Font Arial,Bold is not embedded. Font Arial,Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Italic is not embedded. Font Arial, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed


- (X) Font Arial,Bold is not embedded. Font Arial,Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed 28 more not displayed


- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Italic is not embedded. Font Arial, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Italic is not embedded. Font Arial, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed


- (X) Font Arial,Bold is not embedded. Font Arial,Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed 4 more not displayed

# Page 7 Results

- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed


- (X) Font Arial,Bold is not embedded. Font Arial,Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Italic is not embedded. Font Arial, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed


- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed 5 more not displayed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed 26 more not displayed


- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed


- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed 11 more not displayed